CLINICAL TRIAL: NCT04432857
Title: An Open-Label Multicenter Phase Ib Study of AN0025 in Combination With Pembrolizumab in Patients With Advanced Solid Tumors
Brief Title: AN0025 and Pembrolizumab Combination in Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Adlai Nortye Biopharma Co., Ltd. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AN0025S0103; 2019-003960-37 (EudraCT Number); KEYNOTE-879 (Other: Merck Sharp & Dohme LLC); MK-3475-879 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Triple-negative Breast Cancer; NSCLC, Squamous or Non-Squamous; Urothelial Carcinoma of the Bladder; Microsatellite Stable (MSS) Colorectal Cancer (CRC); Cervical Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Spinocerebellar Degenerations; Colorectal Neoplasms; Uterine Cervical Neoplasms | interventions — E7046; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Ph1a: Urothelial carcinoma of the bladder and NSCLC (Experimental): Patients will receive AN0025 orally once daily (QD); Pembrolizumab, 200mg as an intravenous infusion over 30 minutes every 3 weeks.
  Interventions: Drug: AN0025; Drug: Pembrolizumab
- Phase 1b: Urothelial carcinoma of the bladder (Experimental): Patients will receive AN0025 orally once daily (QD); Pembrolizumab, 200mg as an intravenous infusion over 30 minutes every 3 weeks.
  Interventions: Drug: AN0025; Drug: Pembrolizumab
- Phase 1b: Non-Small Cell Lung Cancer (NSCLC) (Experimental): Patients will receive AN0025 orally once daily (QD); Pembrolizumab, 200mg as an intravenous infusion over 30 minutes every 3 weeks.
  Interventions: Drug: AN0025; Drug: Pembrolizumab
- Phase 1b: Triple-negative breast cancer (TNBC) (Experimental): Patients will receive AN0025 orally once daily (QD); Pembrolizumab, 200mg as an intravenous infusion over 30 minutes every 3 weeks.
  Interventions: Drug: AN0025; Drug: Pembrolizumab
- Phase 1b: Cervical (Experimental): Patients will receive AN0025 orally once daily (QD); Pembrolizumab, 200mg as an intravenous infusion over 30 minutes every 3 weeks.
  Interventions: Drug: AN0025; Drug: Pembrolizumab
- Phase 1b: Microsatellite Stable (MSS) Colorectal Cancer (CRC) (Experimental): Patients will receive AN0025 orally once daily (QD); Pembrolizumab, 200mg as an intravenous infusion over 30 minutes every 3 weeks.
  Interventions: Drug: AN0025; Drug: Pembrolizumab

INTERVENTIONS:
Drug: AN0025 — oral administration
  Other Names: E7046
Drug: Pembrolizumab — Infusion
  Other Names: KEYTRUDA®; MK-3475-879

SUMMARY:
This is an open-label, multicenter, phase Ib study to evaluate the safety and preliminary efficacy of AN0025 in combination with pembrolizumab in patients with locally advanced/metastatic tumors. It will include a dose-limiting toxicity observation phase followed by an expansion phase. All enrolled patients will be treated with AN0025 and Pembrolizumab until the patient experiences disease progression, unacceptable toxicity or withdraws consent, or for a maximum of 35 cycles (approximately 2 years). The dose of pembrolizumab will remain constant at 200 mg every 3 weeks (Q3W) for each dose level of AN0025 and in each cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of informed consent.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
3. Life expectancy ≥3 months.
4. Diagnosed with histologically confirmed locally advanced and nonresectable, or metastatic disease.

   Patients diagnosed with one of the following tumor types:

   A. Urothelial carcinoma of the bladder B. NSCLC, Squamous or Non-Squamous C. TNBC D. Cervical cancer E. MSS CRC
5. Have progressed on treatment with an anti-PD-1/PD-L1monoclonal antibody (mAb) administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies (cohort A, B or C) and have failed available standard of care treatment or deemed inappropriate candidates for additional standard treatments by the investigator. PD-1 treatment progression is defined by meeting all of the following criteria:

   For cohort A, B and C:
   1. Has received at least 2 doses of an approved anti-PD-1/PD-L1 mAb.
   2. Has demonstrated disease progression after PD-1/PD-L1 as defined by RECIST v1.1. The initial evidence of disease progression (PD) is to be confirmed by a second assessment no less than four weeks from the date of the first documented PD, in the absence of rapid clinical progression. i,ii
   3. Progressive disease has been documented within 12 weeks from the last dose of anti-PD-1/L1 mAb.

   i. Seymour et al; iRECIST: Guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol 18: e143-52 ii. This determination is made by the investigator. Once PD is confirmed, the initial date of PD documentation will be considered the date of disease progression.

   For cohort B (NSCLC):
   1. Prior treatments must include an anti-PD-1/PD-L1 mAb AND a platinum-based chemotherapy.
   2. Must include anti-PD-1/PD-L1 mAb or platinum-based chemotherapy was used in one of the following settings:

      * Locally advanced and unresectable
      * Metastatic disease
      * Adjuvant setting with disease progression occurred within 6 months after the last dose
   3. Must include anti-PD-1/PD-L1 mAb or platinum-based chemotherapy was used in one of the following settings:

      * Locally advanced and unresectable
      * Metastatic disease
      * Adjuvant setting with disease progression occurred within 6 months after the last dose or with no prior anti-PD-1/PD-L1 therapy and failed standard of care treatment (cohorts C, D, or E).
6. For cohorts A, C, D and E: Have received no more than 3 prior lines of systemic therapy for advanced disease. Prior therapy in an adjuvant or neoadjuvant setting is not considered as a prior line of systemic therapy. For cohort B (NSCLC), there is no limitation to the number of prior lines of systemic therapy.
7. Have measurable disease per RECIST 1.1 as assessed by the local site investigator and/or radiologist. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
8. Have provided signed informed consent for the trial
9. Have provided archival tumor tissue sample obtained after anti-PD-1/PD-L1 or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
10. Left ventricular ejection fraction (LVEF) greater than 50% on echocardiography or multiple gated acquisition (MUGA) scan.
11. Have adequate organ function.
12. Willing and able to comply with all aspects of the protocol
13. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    1. Not a woman of childbearing potential Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks prior to Screening. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of child-bearing potential.
    2. Woman of childbearing potential who agrees to follow contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.

    Highly effective contraception is defined as either:
    * Total abstinence: When this is in line with the preferred and usual lifestyle of the patient. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
    * Female sterilization: When the female study patient has had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment.
    * Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female study patients, the vasectomized male partner should be the sole partner for that patient.
    * Using a combination of any two of the following:

      * Placement of an intrauterine device (IUD) or intrauterine system (IUS), and
      * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.
      * Hormonal contraception methods (e.g., oral, injected, implanted).
14. A male participant must agree to use contraception during the treatment period and for at least 120 days after the last dose of study treatment.

Exclusion Criteria:

1. Have been discontinued treatment due to a Grade 3 or higher immune-related (irAE) from prior anti-PD-1or anti-PD-L1, or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137)
2. Have received prior systemic anti-cancer therapy including investigational agents within 4 weeks or 5 half-lives, whichever is shorter prior to treatment.

   Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or returned to baseline. Participants with ≤Grade 2 neuropathy may be eligible.
3. Have received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
4. Have received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed. Non live COVID vaccinations or boosters should not occur during Cycle 1 or within 30 days prior to the first dose of study drug.
5. Are currently participating in or have participated in a study of an investigational agent or have used an investigational device within 4 weeks prior to the first dose of study treatment.

   Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been at least 4 weeks after the last dose of the previous investigational agent.
6. Have had an allogenic tissue/solid organ transplant.
7. Have a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. With a history of another primary malignancy within the past 2 years, with the exception of basal or squamous cell skin cancer, or carcinoma in situ of the cervix or breast that has undergone potentially curative therapy.
9. Have known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
10. Have known severe hypersensitivity to study treatment components.
11. Have an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
12. Participants with inflammatory bowel disease.
13. Have a history of (non-infectious) pneumonitis that required steroids or have current pneumonitis.
14. Have an active infection requiring systemic therapy.
15. Participants with known human immunodeficiency virus (HIV) and/or history of Hepatitis B or C infections, or known to be positive for Hepatitis B antigen (HBsAg)/ Hepatitis B virus (HBV) DNA or Hepatitis C Antibody or RNA. Active Hepatitis C is defined by a known positive Hep C Ab result and known quantitative HCV RNA results greater than the lower limits of detection of the assay.
16. Prolongation of corrected QT [QTcF (Fridericia's corrected QT interval)] interval to greater than 480 msec when electrolytes balance is normal.
17. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke within 6 months of the first dose of study drug; or cardiac arrhythmia requiring medical treatment (including oral anticoagulation).
18. Major surgery within 4 weeks before the first dose of study drug. Note: If a participant received major surgery, they must have recovered adequately from surgery and the toxicity and/or complications requiring the intervention prior to starting study treatment.
19. Inability to take oral medication, or malabsorption syndrome or any other uncontrolled gastrointestinal condition (eg, nausea, diarrhea, or vomiting) that might impair the bioavailability of AN0025.
20. Have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
21. Have a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
22. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 3 weeks
  Number of participants with Dose Limiting Toxicities (DLTs)

SECONDARY OUTCOMES:
ORR and Progression-Free Survival (PFS) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 | 2 years
Duration of Response (DOR) | 2 years
Overall Survival (OS) | 2 years
Efficacy by PD-L1 expression | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Atkinson, Ph.D., Study Director — Adlai Nortye US Inc
Locations (6):
- United States (4):
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah School of Medicine Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia, Richmond, Virginia
- France (2):
  - Centre Léon Bérard, Lyon
  - Gustave Roussy, Paris

IPD SHARING:
Plan to Share IPD: No